CLINICAL TRIAL: NCT06415318
Title: A Single-center, Single-arm Clinical Study of TIP(Paclitaxel + Ifosfamide + Cisplatin) Regimen Combined With Triplizumab Neoadjuvant Therapy for Locally Advanced Penile Cancer
Brief Title: TIP Regimen Combined With Triplizumab Neoadjuvant Therapy for Locally Advanced Penile Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Director, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-043-01
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Penile Cancer
MeSH Terms: conditions — Penile Neoplasms | interventions — Paclitaxel; Ifosfamide; Cisplatin; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Neoadjuvant Therapy TIP (Paclitaxel + Ifosfamide + Cisplatin) & Toripalimab (Experimental): Drug: Toripalimab 240mg, ivgtt, d1 Drug: Paclitaxel 175 mg/m2, ivgtt, d1 Drug: Cisplatin 25mg/m2·d, ivgtt, d1-3 Drug: Ifosfamide 1.2g/m2·d, ivgtt, d1-3
  Interventions: Drug: Paclitaxel + Ifosfamide + Cisplatin & Toripalimab

INTERVENTIONS:
Drug: Paclitaxel + Ifosfamide + Cisplatin & Toripalimab — Paclitaxel + Ifosfamide + Cisplatin & Toripalimab

SUMMARY:
Primary Objective: To evaluate the efficacy and safety of TIP (paclitaxel + ifosfamide + cisplatin) combined with Toripalimab as a neoadjuvant treatment in locally advanced penile cancer

DETAILED DESCRIPTION:
Penile cancer is a rare malignant tumor, which often occurs in the inner plate of the prepuce and glans. Squamous cell carcinoma is the most common pathological type. Lymph node metastasis is a crucial factor that leads to poor prognosis of penile cancer. The 5-year OS of penile cancer patients without lymph node metastasis is 90%. Still, it goes down sharply in patients with inguinal lymph node metastasis and pelvic lymph node metastasis, which is 50% and 0%, respectively. Using neoadjuvant chemotherapy to treat patients with locally advanced penile cancer (T4, any N stage, or any T stage, N3) may improve their prognosis. TIP (Paclitaxel + Ifosfamide + Cisplatin) regimen is the first-line neoadjuvant treatment recommended by NCCN guidelines. PD-1 is an immune checkpoint molecule on the surface of T cells. In recent years, immune checkpoint inhibitors targeting PD-1 have shown good efficacy in a variety of tumors. Some phase II / III clinical trials have shown that PD-1 inhibitors can improve the prognosis of patients with lung squamous cell carcinoma, head and neck squamous cell carcinoma, and cervical cancer. Previous studies have found that PD-L1 is highly expressed in 40% - 60% of penile cancer, suggesting that penile cancer patients may benefit from immunotherapy. The management of penile cancer with lymph node metastasis is difficult, especially for the N2-3 stage. This phase II study aims to explore an effective combination therapy for locally advanced penile cancer. 25 patients need to be enrolled.TIP & toripalimab will be administered every 21 days until surgery, evidence of disease progression, or onset of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Squamous cell carcinoma confirmed by histology or cytology;
2. Clinical Stage is Locally advanced penile cancer (T4, any N stage; or any T stage, N3);
3. No prior chemotherapy for newly diagnosed or relapsed patients or the time from the last chemotherapy to relapse should be longer than 12 months;
4. There is at least one measurable lesion according to the solid tumor efficacy evaluation standard RECIST1.1;
5. the Eastern Cooperative Oncology Group (ECOG) scored 0-2;
6. Blood marrow function: Hemoglobin(Hb) >/= 80g/L; White blood cell count >/= 3.0x10^9/L; Neutrophil count >/= 1.5x10^9/L; Platelet count >/ = 100x10^9/L;
7. Liver function: AST, ALT, ALP </= 2.5 ULN; Total bilirubin </= 1.5 ULN;
8. Estimated survival >/= 12 months;
9. No prior serious disease history of a systemic organ;
10. The participant understands this study procedure and signs the informed consent.

Exclusion Criteria:

1. Peripheral neuropathy degree >/=2 (affecting patient's function);
2. Previously received any other experimental drug treatment within 4 weeks before enrollment;
3. Patients with other cancer at present, or have other malignant tumor histories within the past 5 years. Except for (1) Cured skin non-malignant melanoma; (2) Curable tumor, including low-risk prostate cancer (T1a, Gleason score<6, PSA<0.5ng/ml), superficial bladder cancer and so on; (3) Other solid tumors have received radical treatment, and no recurrence or metastasis has been found at least 5 years;
4. Other serious or poorly controlled concomitant diseases, including but not limited to (1) Severe or acute attack disease history of cardiovascular, liver, respiratory, kidney, blood, endocrine or neuropsychiatric system within 6 months; (2) Active infection history and needed antibiotic treatment within 2 weeks before enrollment; (3) Congestive heart failure (grade III-IV); (4) Unstable angina pectoris or myocardial infarction history within 6 months

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 weeks
  Objective Response Rate (ORR) based on RECIST 1.1 criteria.

SECONDARY OUTCOMES:
pCR | 12 weeks
  Percentage of Participants With Pathologically Complete Response
EFS | 2 months
  Event-free survival, EFS
OS | 6 months
  Overall Survival
Adverse events | 2 months
  Number of participants with treatment-related adverse events as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No